CLINICAL TRIAL: NCT05287464
Title: International Multicentric Study ARON-1
Status: Recruiting | Type: Observational
Sponsor: Hospital of Macerata (Other)
Responsible Party: Sponsor
Other Study IDs: ARON-1
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Renal Cell Carcinoma (mRCC)
Keywords: immunotherapy; mRCC; immuno-combinations; artificial intelligence technology; real-world data
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; Axitinib; Nivolumab; cabozantinib; lenvatinib; Ipilimumab; avelumab; atezolizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: pembrolizumab plus axitinib — collect global experiences with the use of immuno-combinations in patients with metastatic RCC
  Other Names: nivolumab plus cabozantinib; pembrolizumab plus lenvatinib; nivolumab plus ipilimumab; avelumab plus axitinib; atezolizumab plus bevacizumab

SUMMARY:
The ARON-1 Study is designed as an International Multicentric Retrospective Study to collect global experiences with the use of immuno-combinations in patients with metastatic RCC.

Two Supplementary Studies (ARON-1α and ARON-1β) have been designed. The ARON-1α Supplementary Study has been designed to investigate for the presence of genomic signatures from tumor samples of patients treated with first-line immuno-combinations for advanced RCC. The ARON-1β Supplementary Study has been designed to charaterize the immune cell populations and assess their relationship with the clinical outcome of mRCC patients treated with first-line immuno-combinations

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18y
* Cytological or Histologically confirmed diagnosis of clear cell or non-clear cell RCC
* Histologically or radiologically confirmed diagnosis of metastatic disease
* First-line treatment with nivolumab plus ipilimumab or nivolumab plus cabozantinib or pembrolizumab plus axitinib or pembrolizumab plus lenvatinib or avelumab plus axitinib or atezolizumab plus bevacizumab

Exclusion Criteria:

* Patients without histologically confirmed diagnosis of RCC
* Patients without histologically or radiologically confirmed metastatic disease
* Patients treated with immuno-combinations not included in the list reported in the Inclusion Criteria Section

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with first-line immuno-combinations for metastatic RCC
Sampling Method: Probability Sample
Enrollment: 1220 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | March 31th, 2022
Overall Survival (OS) | March 31th, 2022
Overall Response Rate (ORR) | March 31th, 2022

SECONDARY OUTCOMES:
Efficacy of immuno-combination in the elderly populaton | May 31th, 2022
  Data on tumor assessment and response to therapy on elderly populaton will be statistically analyzed
Efficacy of immuno-combinations in patients with different metastatic sites (i.e. bone and brain metastases) | May 31th, 2022
  Data on tumor assessment and response to therapy will be statistically analyzed
Prognostic role of smoking attitude and obesity in RCC patients treated with different immuno-combinations | May 31th, 2022
  Statistical analysis of prognostic role of smoking attitude and obesity in treated RCC patients
Efficacy of different immuno-combinations in patients with non-clear RCC | September 30th, 2022
  Data on tumor assessment and response to therapy in non-clear RCC will be statistically analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale di Macerata, UOC Oncologia, Macerata, Macerata, Italy

REFERENCES:
- [Derived] Santoni M, Massari F, Myint ZW, Iacovelli R, Pichler M, Basso U, Kopecky J, Kucharz J, Buti S, Rizzo M, Galli L, Buttner T, De Giorgi U, Kanesvaran R, Fiala O, Grande E, Zucali PA, Fornarini G, Bourlon MT, Scagliarini S, Molina-Cerrillo J, Aurilio G, Matrana MR, Pichler R, Cattrini C, Buchler T, Seront E, Calabro F, Pinto A, Berardi R, Zgura A, Mammone G, Ansari J, Atzori F, Chiari R, Bamias A, Caffo O, Procopio G, Bassanelli M, Merler S, Messina C, Kuronya Z, Mosca A, Bhuva D, Vau N, Incorvaia L, Rebuzzi SE, Roviello G, Zabalza IO, Rizzo A, Mollica V, Sorgentoni G, Monteiro FSM, Montironi R, Battelli N, Porta C. Global Real-World Outcomes of Patients Receiving Immuno-Oncology Combinations for Advanced Renal Cell Carcinoma: The ARON-1 Study. Target Oncol. 2023 Jul;18(4):559-570. doi: 10.1007/s11523-023-00978-2. Epub 2023 Jun 27. PMID 37369815
- [Derived] Santoni M, Massari F, Myint ZW, Iacovelli R, Pichler M, Basso U, Kopecky J, Kucharz J, Buti S, Salfi A, Buttner T, De Giorgi U, Kanesvaran R, Fiala O, Grande E, Zucali PA, Fornarini G, Bourlon MT, Scagliarini S, Molina-Cerrillo J, Aurilio G, Matrana MR, Pichler R, Cattrini C, Buchler T, Seront E, Calabro F, Pinto A, Berardi R, Zgura A, Mammone G, Ansari J, Atzori F, Chiari R, Zakopoulou R, Caffo O, Procopio G, Bassanelli M, Zampiva I, Messina C, Kuronya Z, Mosca A, Bhuva D, Vau N, Incorvaia L, Rebuzzi SE, Roviello G, Zabalza IO, Rizzo A, Mollica V, Catalini I, Monteiro FSM, Montironi R, Battelli N, Rizzo M, Porta C. Clinico-Pathological Features Influencing the Prognostic Role of Body Mass Index in Patients With Advanced Renal Cell Carcinoma Treated by Immuno-Oncology Combinations (ARON-1). Clin Genitourin Cancer. 2023 Oct;21(5):e309-e319.e1. doi: 10.1016/j.clgc.2023.03.006. Epub 2023 Mar 20. PMID 37062658